CLINICAL TRIAL: NCT05976685
Title: Early Closure of Left Atrial Appendage for Patients With Atrial Fibrillation and Ischemic StrokE Despite Anticoagulation Therapy
Acronym: ELAPSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-02340
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Stroke; Atrial Fibrillation
Keywords: Stroke; Direct oral anticoagulation; Left atrial appendage occlusion
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation; Stroke | interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LAAO and DOAC therapy (Experimental): Left atrial appendage occlusion and therapy with direct oral anticoagulants
  Interventions: Procedure: Left atrial appendage Occlusion; Drug: DOAC
- DOAC therapy only (Other): Therapy with direct oral anticoagulants alone
  Interventions: Drug: DOAC

INTERVENTIONS:
Procedure: Left atrial appendage Occlusion — Left atrial appendage Occlusion and therapy with direct oral anticoagulants. Choice of DOAC is at the discretion of the treating physician.
  Arms: LAAO and DOAC therapy
Drug: DOAC — Therapy with direct oral anticoagulants. Choice of DOAC is at the discretion of the treating physician.

SUMMARY:
Atrial fibrillation (AF) is one of the most common cardiac arrhythmias and cardioembolic stroke due to AF is its major complication. Direct oral anticoagulants (DOAC) reduce the risk of cardioembolism in patients with AF. Despite DOAC therapy, there is a significant residual stroke risk of 1-2%/year. Recent data from the Swiss Stroke Registry found 38% of patients with AF and ischemic stroke were on prior anticoagulant therapy (approximately 400 patients per year in Switzerland). The investigators found in a prior observational study, that patients with AF who have ischemic stroke despite anticoagulation are at increased risk of having another ischemic stroke (HR 1.6; 95% confidence interval, CI 1.1-2.1). Combining observational data from 11 international stroke centres, the investigators found that the majority of ischemic strokes despite anticoagulation in patients with AF is "breakthrough" cardioembolism (76% of patients) and only a minority of 24% is related to other causes unrelated to AF. Optimal secondary prevention strategy is unknown. The investigators have conducted two independent observational studies including together >4000 patients but did not identify any strategy (e.g. switch to different DOAC, additional antiplatelet therapy) that seems superior. A recent randomized controlled trial on surgical occlusion of the left atrial appendage (LAAO) found that LAAO may provide additional protection from ischaemic stroke in addition to oral anticoagulation. Triggered by this finding, the investigators performed a matched retrospective observational study and found that patients with AF and stroke despite anticoagulation who received a combined mechanical-pharmacological therapy (DOAC therapy + LAAO) had lower rates of adverse outcomes compared to those with DOAC therapy alone. Therefore, the investigators hypothesize that in patients with AF and ischemic stroke despite anticoagulant therapy, LAAO in addition to anticoagulation with a DOAC is superior to DOAC therapy alone. The investigators propose an international, multi-center randomized controlled two-arm trial to assess the effect of LAAO in patients with AF suffering from strokes despite anticoagulation therapy and without competing stroke etiology. The investigators will use the PROBE design with blinded endpoint assessment. The investigators will enrol patients with non-valvular AF and a recent ischemic stroke despite anticoagulation therapy at stroke onset. Patients will be randomized 1:1 to receive LAAO + DOAC therapy (experimental arm) or DOAC therapy alone (standard treatment arm). The primary endpoint is the first occurrence of a composite outcome of recurrent ischemic stroke, systemic embolism and cardiovascular death during follow-up. Secondary outcomes include individual components of the primary composite outcome, safety outcomes (i.e. symptomatic intracranial haemorrhage, major extracranial bleeding, serious device- or procedure-related complication), functional outcome (modified Rankin Scale) and patient-oriented outcomes. The minimum follow-up is 6 months and all patients will receive follow-ups every 6 months until end of study, the maximal follow-up will be 48 months. Based on prior observational data from the investigators' group and others (5 observational studies, >5000 patients), the investigators estimate the proportion of patients with the primary outcome in the standard treatment arm to be 18% in the first year and 9% in the second year (=cumulative 27% after 2 years). A relative risk reduction of 40% at 2 years would be clinically relevant. Based on these assumptions and a log-rank test, the investigators would need 98 events for a power of 80% at an alpha-level of 5%. Assuming a recruitment rate of 52, 118, 156 and 156 patients in years 1 to 4, an additional 6 months of follow-up (mean follow-up time of 2.1 years) and a uniform drop-out rate of 7.5% per year, 482 patients would need to be enrolled. How to treat patients with an ischemic stroke despite anticoagulation is a major yet unresolved clinical dilemma. This trial has the potential to answer the question whether LAAO plus DOAC therapy is superior to current standard of care for patients with AF who have ischemic stroke despite anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Written informed consent
* Permanent, persistent, or paroxysmal spontaneous AF previously known or diagnosed during the index hospitalization.
* Recent (≤3 months) symptomatic ischemic stroke.
* Active and ongoing anticoagulation therapy at stroke onset assessed based on medical history (i.e. any therapeutic oral anticoagulation therapy [Vitamin K antagonist/DOAC according to prescription recommendations for AF; inadequate low-dose DOAC therapy allowed for inclusion] not stopped/paused for >48 hours due to any reason, i.e. medical intervention or non-adherence).
* Active or planned long-term therapy with DOAC

Exclusion Criteria:

* Contraindications to DOAC therapy
* Life expectancy <1 year according to the opinion of the investigator
* Stroke due to: Ipsilateral intra/extracranial high-grade stenosis, Isolated lacunar stroke, Other well-defined stroke aetiologies (i.e., endocarditis, vasculitis, Reversible Cerebral Vasoconstriction Syndrome [RCVS], Posterior Reversible Encephalopathy Syndrome [PRES], cerebral sinus venous thrombosis)
* Previous persistent foramen ovale or atrial septum defect closure.
* Rheumatic heart disease
* Severe heart valve disease that requires treatment (severe aortic stenosis or regurgitation, severe mitral stenosis or regurgitation).
* Contraindications for TEE (relevant esophageal varices, esophageal stricture, history of esophageal cancer).
* Cardiac or non-cardiac surgical procedure within 30 days of randomization
* Enrolled in another investigation of a cardiovascular device or investigating secondary prevention therapy.
* Severely reduced Left Ventricular Ejection Fraction (LVEF) <30%.
* Severe renal impairment as described in the summary of medicinal product characteristics for the chosen DOAC (e.g. rivaroxaban, apixaban and edoxaban creatinine clearance <15 ml/min; dabigatran creatinine clearance <30 ml/min).
* Hypertrophic cardiomyopathy
* Intracardiac tumor
* Ventricular thrombus
* Acute cardiac decompensation
* LAA is obliterated or surgically ligated
* Persistent proximal LAA thrombus despite 4 weeks of anticoagulation (if a proximal thrombus in the LAA is found, anticoagulation with vitamin K antagonist (INR 2.5-3.5) may be started, and if the thrombus disappears, the patient may be eligible for LAAO)
* Pregnancy or breastfeeding (pregnancy test in urine or blood to be performed at screening for women of childbearing potential)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 482 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Composite of recurrent ischemic stroke, systemic embolism, or cardiovascular death (whatever comes first). | 6 months
  The primary endpoint is the first occurrence of a composite outcome of recurrent ischemic stroke, systemic embolism and cardiovascular death during follow-up. Stoke is defined as - New sudden focal neurological deficit of presumed cerebrovascular aetiology, occurring > 24 hours after the index ischaemic stroke, that persisted beyond 24 hours and was not due to another identifiable cause 18 (transient ischaemic attack (TIA), defined as a transient episode of neurologic dysfunction caused by focal brain, spinal cord, or retinal ischaemia without cerebral infarction on imaging, is not judged as stroke) and/or by brain imaging (CT or MRI). Systemic embolism is defined as abrupt vascular insufficiency associated with clinical or radiological evidence of arterial occlusion of an extremity or organ in absence of another likely mechanism (e.g. atherosclerosis, instrumentation or trauma). Cardiovascular death is defined as any death that is due to a vascular cause.

SECONDARY OUTCOMES:
Recurrent ischemic stroke | 6 months
  Stoke is defined as - New sudden focal neurological deficit of presumed cerebrovascular aetiology, occurring > 24 hours after the index ischaemic stroke, that persisted beyond 24 hours and was not due to another identifiable cause 18 (transient ischaemic attack (TIA), defined as a transient episode of neurologic dysfunction caused by focal brain, spinal cord, or retinal ischaemia without cerebral infarction on imaging, is not judged as stroke) and/or by brain imaging (CT or MRI).
Systemic embolism | 6 months
  Systemic embolism is defined as abrupt vascular insufficiency associated with clinical or radiological evidence of arterial occlusion of an extremity or organ in absence of another likely mechanism (e.g. atherosclerosis, instrumentation or trauma).
Cardiovascular death | 6 months
  Cardiovascular death is defined as any death that is due to a vascular cause.
Symptomatic intracranial hemorrhage | 6 months
  A relevant symptomatic intracranial haemorrhage, this includes subdural, epidural, subarachnoidal and intracerebral haemorrhage, is defined as haemorrhage that leads to a clinical worsening and hospitalisation and is assessed by the treating physician to be likely the cause of the new neurological symptom or the death. Intracerebral haemorrhage due to a trauma will not be considered.
Major extracranial bleeding (ISTH) | 6 months
  Definition released by the International Society of Thrombosis and Haemostasis (ISTH): clinically overt bleeding which was fatal or associated with any of the following: (a) a fall in hemoglobin level of 2 g/dL or more or documented transfusion of at least 2 units of packed red blood cells, (b) involvement of a critical anatomical site (intracranial, spinal, ocular, pericardial, articular, intramuscular with compartment syndrome, retroperitoneal).
Procedure-related death | 6 months
  All-cause death within 30 days after randomization or during the index procedure hospitalization
Serious device- or procedure-related complication | 6 months
  7 days post-index procedure for device group subjects
All-cause hospitalization | 6 months
  Any hospital stay of at least 24 hours
Cause-specific hospitalization | 6 months
  Any hospital stay of at least 24 hours or which the primary admitting diagnosis was for heart failure, stroke, bleeding, atrial fibrillation, repeat AF-ablations, periprocedural complication, other cardiovascular causes
Global health | 6 months
  Measured by PROMIS (Patient-reported Outcomes Measurement Information System) Adult Global Health; continuous
Global safety | 6 months
  Measured by FeelSaveScale; continuous
Functional neurological outcome | 6 months
  Modified Rankin Scale; ordinal

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Räber, Prof., MD, Principal Investigator — Cardiovascular Center, Inselspital Bern
Locations (23):
- Belgium (5):
  - AZ Sint Jan Brugge, Bruges
  - Brussels University Hospital, Brussels
  - UCLouvain - Cliniques universitaires Saint-Luc, Brussels
  - HUmani CHU Charleroi-Chimay, Charleroi
  - Universitair Ziekenhuis (UZ) Leuven, Leuven
- Germany (8):
  - UKSH, Campus Lübeck, Lübeck, Schleswig-Holstein
  - Charité-Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Universitätsmedizin Göttingen, Göttingen
  - Asklepios Klinik Altona, Hamburg
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsmedizin Mannheim, Mannheim
  - Universitätsklinikum Tübingen, Tübingen
- Christchurch Hospital, Christchurch, New Zealand
- Switzerland (7):
  - Ente Ospedaliero Cantonale, Lugano, Canton Ticino
  - Centre Hospitalier Universitaire Vaudois, Lausanne, Vaude
  - University Hospital Basel, Basel
  - Inselspital, University Hospital Bern, Bern
  - Hôpitaux universitaires de Genève, Geneva
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen
- United Kingdom (2):
  - St Thomas' Hospital, London
  - University Hospitals Sessex NHS Trust, Worthing

IPD SHARING:
Plan to Share IPD: No